CLINICAL TRIAL: NCT05628129
Title: Effect of WeChat Application Combined Phone Reminder on Follow-up Adherence Improvement in Congenital Ectopia Lentis Patients : A Randomized Controlled Trial
Brief Title: Effect of Mobile Communication on Congenital Ectopia Lentis Follow-up Adherence
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IIT2022120
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Ectopia Lentis
MeSH Terms: conditions — Ectopia Lentis

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reminder intervention (Experimental): On the basis of standard appointment, parents in intervention group will receive phone reminders at 4 days and 1 day before their scheduled appointments, and relevant scientific and educational knowledge will be relayed to them from the smartphone application at 1 week before appointments.
  Interventions: Other: smartphone application service and phone reminder
- standard appointment (No Intervention): Patients will be required to attend follow-up appointments at 1 week, 1 month, 3 months after surgery.

INTERVENTIONS:
Other: smartphone application service and phone reminder — smartphone application service and phone reminder for appointments of parents of congenital ectopia lentis patients
  Arms: reminder intervention

SUMMARY:
Regular follow-up is essential to successful management of congenital ectopia lentis, but it is often ignored by parents in China.

With rapid economic development, there are increasing numbers of mobile phone users that allow for communication applications to be used in medical care.

The investigators aimed to assess the potential of the smartphone application assisted medical service to increase patient compliance in attendance of follow-up after congenital ectopia lentis treatment.

DETAILED DESCRIPTION:
Congenital ectopia lentis is a rare ophthalmic disease that seriously harms the physical and mental health of patients. Surgery is the only definite treatment at present. However, severe visual impairment is common in congenital ectopia lentis patients in China, and delayed presentation to hospital and late surgical treatment are found to be the major reasons.

In China, the messaging application WeChat has become the most popular communication tool. As most congenital ectopia lentis patients' parents are younger people, they are more likely to use technology, such as WeChat, in their daily lives. In addition, it allows ophthalmologists to utilize this communication application to relay health related information and reminders to patients. This makes it feasible to apply this smartphone application in improving attendance of follow-up visits.

In this trial, the investigators aimed to assess the potential of the smartphone application assisted medical service to increase patient compliance in attendance of follow-up after congenital ectopia lentis treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Identified with congenital lens dislocation after surgery and age ≤ 18 years old; 2. Parents were able to access a mobile phone and communicate via the smartphone application (WeChat); 3. Agree to participate in this study and sign the informed consent.

Exclusion Criteria:

* 1. With Other ophthalmic diseases such as glaucoma, uveitis and corneal disease.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
follow-up adherence at 3 months after surgery | 3 months
  the rates of attendance at 3 months (± 3 weeks) after surgery

SECONDARY OUTCOMES:
follow-up adherence at 1 week after surgery | 1 week
  the rates of attendance at 1 week (± 2 days) after surgery
follow-up adherence at 1 month after surgery | 1 month
  the rates of attendance at 1 month (± 1 week) after surgery
best corrected visual acuity | 3 months
  measurement of best corrected visual acuity was carried out using a logarithm of the Minimum Angle of Resolution (logMAR) chart at the baseline and endline visits
replacement rates of glasses | 3 months
  If the difference between the current refraction and the currently worn eyeglass prescription was greater than 2 diopters sphere and/or greater than 1 diopter cylinder, a new prescription was given
amblyopia therapy rate | 3 months
  the rate of amblyopia therapy during 3 months after surgery
referral rate due to systemic diseases | 3 months
  referral rate due to abnormalities in skeletal system and cardiovascular system during 3 months after surgery
CEL knowledge score | 3 months
  change between baseline and endline scores on knowledge about CEL, including six choice questions concerning pathogenesis, symptoms and treatment of CEL

OTHER OUTCOMES:
follow-up adherence at 6 months after surgery | 6 months
  the rates of attendance at 6 months (± 1 month) after surgery
follow-up adherence at 1 year after surgery | 1 year
  the rates of attendance at 1 year (± 2 months) after surgery
follow-up adherence at 2 years after surgery | 2 years
  the rates of attendance at 2 years (± 4 months) after surgery
follow-up adherence at 3 years after surgery | 3 years
  the rates of attendance at 3 years (± 6 months) after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Danying Zheng, M.D, Principal Investigator — Clinical Research Center of Zhongshan Ophthalmic Center
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin H, Chen W, Luo L, Congdon N, Zhang X, Zhong X, Liu Z, Chen W, Wu C, Zheng D, Deng D, Ye S, Lin Z, Zou X, Liu Y. Effectiveness of a short message reminder in increasing compliance with pediatric cataract treatment: a randomized trial. Ophthalmology. 2012 Dec;119(12):2463-70. doi: 10.1016/j.ophtha.2012.06.046. Epub 2012 Aug 24. PMID 22921386
- [Background] Chen T, Zhu W, Tang B, Jin L, Fu H, Chen Y, Wang C, Zhang G, Wang J, Ye T, Xiao D, Vignarajan J, Xiao B, Kanagasingam Y, Congdon N. A Mobile Phone Informational Reminder to Improve Eye Care Adherence Among Diabetic Patients in Rural China: A Randomized Controlled Trial. Am J Ophthalmol. 2018 Oct;194:54-62. doi: 10.1016/j.ajo.2018.07.006. Epub 2018 Jul 24. PMID 30053472
- [Background] Lin J, Gong N, Cao Q, Zhou Y, Cai Y, Jin G, Young CA, Yang J, Wang Y, Zheng D. What hinders congenital ectopia lentis patients' follow-up visits? A qualitative study. BMJ Open. 2020 Mar 12;10(3):e030434. doi: 10.1136/bmjopen-2019-030434. PMID 32169922
- [Background] Tan J, Christie A, Montalvo SK, Wallace C, Yan Y, Folkerts M, Yingling A, Sher D, Choy H, Jiang S, Westover KD. Automated Text Message Reminders Improve Radiation Therapy Compliance. Int J Radiat Oncol Biol Phys. 2019 Apr 1;103(5):1045-1052. doi: 10.1016/j.ijrobp.2018.11.050. Epub 2018 Nov 30. PMID 30508618
- [Background] Bi J, Yang W, Hao P, Zhao Y, Wei D, Sun Y, Lin Y, Sun M, Chen X, Luo X, Li S, Zhang W, Wang X. WeChat as a Platform for Baduanjin Intervention in Patients With Stable Chronic Obstructive Pulmonary Disease in China: Retrospective Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Feb 2;9(2):e23548. doi: 10.2196/23548. PMID 33528369
- [Background] Yang K, Jin L, Li L, Zeng S, Wei R, Li G, Man P, Congdon N. Interventions to Promote Follow-up After Trabeculectomy Surgery in Rural Southern China: A Randomized Clinical Trial. JAMA Ophthalmol. 2016 Oct 1;134(10):1135-1141. doi: 10.1001/jamaophthalmol.2016.2819. PMID 27541442
- [Derived] Ma Y, Zhang X, Jin L, Liu S, Liang X, Ye Q, Liu X, Congdon N, Zheng D, Jin G. Social Media Interventions and Postoperative Follow-Up in Congenital Ectopia Lentis: A Randomized Clinical Trial. JAMA Ophthalmol. 2025 May 1;143(5):438-445. doi: 10.1001/jamaophthalmol.2025.0526. PMID 40208617